CLINICAL TRIAL: NCT00948220
Title: Non-randomized Prospective Study on the Effect of Antiviral Therapy With Peginterferon Alfa-2a and Ribavirin on Bone Mineral Density and Metabolism in Patients With Chronic Viral Hepatitis C Genotype 1
Brief Title: Influence of Antiviral Therapy on Bone Mineral Density and Metabolism in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. med. D. Klass, Universitätsklinikum Ulm
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OSTEO
Record Dates: First submitted 2009-07-24; First posted 2009-07-29 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-05

CONDITIONS: Hepatitis C, Chronic; Liver Diseases; Virus Diseases
Keywords: HCV; hepatitis C virus; CHC; chronic hepatitis c; interferon; ribavirin; DEXA; BMD; bone mineral density; osteoporosis; osteopenia; osteodystrophy; osteodensitometry; Bone Density; Hepatitis, Viral, Human; Anti-Infective Agents; peginterferon alfa-2a
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Virus Diseases; Hepatitis C; Osteoporosis; Bone Diseases, Metabolic; Hepatitis, Viral, Human | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Chronic hepatitis C patients on standard antiviral therapy with peginterferon alfa-2a and ribavirin
  Interventions: Drug: peginterferon alfa-2a and ribavirin
- Control (No Intervention): Chronic hepatitis C patients without standard antiviral therapy

INTERVENTIONS:
Drug: peginterferon alfa-2a and ribavirin — standard antiviral therapy with peginterferon alfa-2a 180 µg/week and ribavirin 1000-1200 mg/d
  Other Names: Pegasys; Copegus
  Arms: Treatment

SUMMARY:
One single study has suggested that bone mineral density (BMD) is reduced in patients with non-cirrhotic chronic viral hepatitis C. Antiviral combination therapy with standard interferon and ribavirin may further decrease BMD. The aim of this study is to systematically investigate the effect of chronic hepatitis C genotype 1 infection alone and current standard therapy with peginterferon alfa-2a/ribavirin on BMD and bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* proven chronic hepatitis C
* aged between 18 and 65
* male patients

Exclusion Criteria:

* high grade liver fibrosis (Grade 3 - 4)
* renal disease
* hyperparathyroidism
* hypogonadism
* malignant disease
* use of any other drug known to effect bone mineral metabolism
* use of alcohol
* organ transplant
* any form of thyroid disease
* any medical condition known to be associated with bone loss

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-07; Primary Completion 2007-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change of the bone mineral density of the lumbar spine and right hip measured by DEXA in patients with chronic hepatitis C with or without antiviral combination treatment with peginterferon and ribavirin | 96 weeks

SECONDARY OUTCOMES:
Change in markers of bone formation and resorption over time during antiviral therapy and after cessation of therapy. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fuchs, MD, Principal Investigator — University of Ulm
Locations (1):
- University Hospital Ulm, Ulm, Germany